CLINICAL TRIAL: NCT04737369
Title: Multimodal Neuromonitoring: an Explorative Study in Neurocritical Care Patients
Brief Title: Multimodal Neuromonitoring
Acronym: MMNM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Karl Landsteiner Institute for Clinical Epilepsy Research (Other Government)
Responsible Party: Principal Investigator, Johannes Herta, Principle Investigator, Co-Head of the Neurosurgical ICU, Medical University of Vienna
Other Study IDs: MMNM01
Record Dates: First submitted 2020-06-09; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Traumatic Brain Injury; Cortical Spreading Depolarization and Depression; Seizures; Ictal-Interictal Continuum
Keywords: Multimodal Neuromonitoring; Electrocorticography; Cerebral Microdialysis; Neuropharmacology
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Brain Injuries, Traumatic; Depression; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microdialysis Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Theoretical Framework & Background

Cortical spreading depressions (CSD) and seizures, are crucial in the development of delayed cerebral ischemia and poor functional outcome in patients suffering from acute brain injuries such as subarachnoid hemorrhage. Multimodal neuromonitoring (MMNM) provides the unique possibility in the sedated and mechanically ventilated patients to record these electrophysiological phenomena and relate them to measures of cerebral ischemia and malperfusion. MMNM combines invasive (e.g. electrocorticography, cerebral microdialysis, brain tissue oxygenation) and noninvasive (e.g. neuroimaging, continuous EEG) techniques. Additionally, cerebral microdialysis can measure the unbound extracellular drug concentrations of sedatives, which potentially inhibit CSD and seizures in various degrees, beyond the blood-brain barrier without further interventions.

Hypotheses

1. Online multimodal neuromonitoring can accurately detect changes in neuronal metabolic demand and pathological neuronal bioelectrical changes in highly vulnerable brain tissue.
2. Online multimodal neuromonitoring can accurately detect the impact of pathological neuronal bioelectrical changes on metabolic demand in highly vulnerable brain tissue.
3. The occurrence and duration of pathological neuronal bioelectrical changes are dependent on sedatives and antiepileptic drug concentrations
4. The occurrence and duration of pathological neuronal bioelectrical changes have a negative impact on functional and neurological long-term patient outcome.
5. Simultaneous invasive and non-invasive multimodal neuromonitoring can identify a clear relationship of both methods regarding pathological neuronal bioelectrical changes and metabolic brain status.

Methods

Systematic analysis of MMNM measurements following standardized criteria and correlation of electrophysiological phenomena with cerebral metabolic changes in all included patients. In a second step neuroimaging, cerebral extracellular sedative drug concentrations and neurological functional outcome, will be correlated with both electrophysiologic and metabolic changes. Due to numerous high-resolution parameters, machine learning algorithms will be used to correlate comprehensive data on group and individual levels following a holistic approach.

Level of originality

Extensive, cutting edge diagnostic methods are used to get a better insight into the pathophysiology of electrophysiological and metabolic changes during the development of secondary brain damage. Due to the immense amount of high-resolution data, a computer-assisted evaluation will be applied to identify relationships in the development of secondary brain injury. For the first time systematic testing of several drug concentrations beyond the blood-brain barrier will be performed. With these combined methods, we will be able to develop new cerebroprotective treatment concepts on an individual basis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 18-80 years with poor grade aneurysmal SAH (World Federation Neurosurgical Societies >3), severe ICH (ICH Score >3) or severe TBI (Glasgow Coma Scale < 9). The diagnosis of SAH, ICH and TBI will be established by computed tomography (CT).
* Individuals that are unlikely to regain consciousness within the following 48 hours.
* Individuals that are expected to survive for the next 48 hours.

Exclusion Criteria:

* Individuals younger than 18 years old and older than 80 years.
* Pregnant women (documented via positive ß-HCG test).
* Patients, who do not want to participate in the study. As the patient is not able to consent prior to the study, information about the study details will be given to the patient in case of clinical improvement. The patient information sheet will be handed out.

Thereafter, the patient has the possibility to withdraw permission of study-participation.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals between 18-80 years with poor grade aneurysmal SAH (World Federation Neurosurgical Societies >3), severe ICH (ICH Score >3) or severe TBI (Glasgow Coma Scale <9).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Count of SD during electrocorticography | up to 21 days
  Count of cortical spreading depolarization (SD) during continuous electrocorticography
Daily pattern duration of CSD during electrocorticography | up to 21 days
  Duration of cortical spreading depression (CSD) per hour during continuous electrocorticography
Daily pattern duration of NCSE during electrocorticography | up to 21 days
  Duration of nonconvulsive status epilepticus (NCSE) per hour during continuous electrocorticography
Daily pattern duration of RPPIIC during electrocorticography | up to 21 days
  Duration of rhythmic or periodic EEG patterns on the ictal-interictal continuum (RPPIIC) per hour during continuous electrocorticography
Daily duration of metabolic crisis | up to 21 days
  Duration of metabolic crisis (defined as Lactate Pyruvate ratio [LPR] > 40 and lactate higher than 4 mmol/l) during continuous electrocorticography
Daily duration of mitochondrial dysfunction | up to 21 days
  Duration of mitochondrial dysfunction (defined as LPR > 40, Pyruvate > 70 μmol/l and partial brain tissue oxygenation [PbtO2] > 20 mmHg) during continuous electrocorticography
Daily duration of ischemia | up to 21 days
  Duration of ischemia (defined as PbtO2 < 15 mmHg and cerebral perfusion pressure [CPP] < 60 mmHg) during continuous electrocorticography
Daily duration of elevated intracranial pressure (ICP) | up to 21 days
  Duration of elevated intracranial pressure (defined as ICP > 22 mmHg) during continuous electrocorticography
Neuropharmacology Cmax) | up to 21 days
  Cmax of routinely used sedative drug concentrations in blood and brain (Esketamine, Midazolam and Propofol)
Neuropharmacology (AUC) | up to 21 days
  AUC of routinely used sedative drug concentrations in blood and brain (Esketamine, Midazolam and Propofol)
Neuropharmacology (t1/2) | up to 21 days
  t1/2 of routinely used sedative drug concentrations in blood and brain (Esketamine, Midazolam and Propofol)
Neuroimaging | up to 28 days
  Absence or presence of hypoperfusion or ischemic infarctions in neuroimaging
Functional patient outcome | up to 6 months
  modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Herta, MD PhD, Principal Investigator — Department of Neurosurgery, Medical University of Vienna
Locations (1):
- Department of Neurosurgery, Medical University of Vienna, Vienna, Austria